CLINICAL TRIAL: NCT07406113
Title: MEOP - Multidimensional Evaluations in Oncological Psychiatry
Acronym: MEOP
Status: Not yet recruiting | Type: Observational
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Sponsor
Other Study IDs: 7944
Record Dates: First submitted 2026-01-15; First posted 2026-02-12 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-01

CONDITIONS: Psychiatric Disorder; Cognition Disorder; Treatment Compliance; Adverse Drug Event; Family Members
MeSH Terms: conditions — Mental Disorders; Cognition Disorders; Patient Compliance; Drug-Related Side Effects and Adverse Reactions | interventions — Psychiatry; Hematologic Tests

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (6):
- Cases: any subject affected by cancer with a comorbid psychiatric disorder
  Interventions: Behavioral: Psychiatric and neuropsychological evaluation through rating scales
- cases-rel: any first-degree relative of a subject of a "case" (i.e., i.e. a fist-degree relative of a subject affected by cancer and a psychiatric disorder
  Interventions: Behavioral: Psychiatric and neuropsychological evaluation through rating scales
- oncology-controls: Subjects with cancer who will undergo a consultation in the Clinical and Emergency Psychiatry Unit of the Fondazione Policlinico Universitario Agostino Gemelli IRCCS but who do not show any psychiatric symptoms
  Interventions: Behavioral: Psychiatric and neuropsychological evaluation through rating scales
- psy-controls: subjects without cancer who will undergo a psychiatric evaluation in the Clinical and Emergency Psychiatry Unit and present psychiatric symptoms
  Interventions: Behavioral: Psychiatric and neuropsychological evaluation through rating scales
- healthy controls: Subjects without cancer and with any suspected psychiatric disorder who will undergo a psychiatric evaluation in the Clinical and Emergency Psychiatry Unit and who are not diagnosed with any relevant psychiatric symptoms after the evaluation
  Interventions: Behavioral: Psychiatric and neuropsychological evaluation through rating scales
- control-rel: First-degree relatives of "oncology-controls", "psy-controls" and "healthy controls"
  Interventions: Behavioral: Psychiatric and neuropsychological evaluation through rating scales

INTERVENTIONS:
Behavioral: Psychiatric and neuropsychological evaluation through rating scales — Psychiatric evaluation: a) assessment of previous psychiatric history and family history; b) assessment of the presence of a psychiatric syndrome;c) evaluation of mental status; d) evaluation and documentation of psychopharmacological and psychotherapeutic treatments assumed; e) documentation of any side effects related to treatment.
  Administration of psychiatric rating scales. Clinical evaluation: a) collection of medical history; b) recording of chemo- or radiotherapy assumed and current pharmacological treatments; c) physical examination.
  Blood samples Neuropsychological evaluation that will include a series of tests investigating different neurocognitive domains.
  Other Names: Medical evaluation and blood testing.

SUMMARY:
Cancer is among the leading causes of morbidity and mortality worldwide, profoundly affecting patients' lives at every level, and its psychological and psychiatric impacts remain a major concern. Psychiatric disorders are frequently observed in cancer patients. Nevertheless, they were also underdiagnosed, with a consequent undermining possible interventions. Still, psychiatric disorders in cancer patients are not merely secondary complications but may actively contribute to poor oncological outcomes.

The pathophysiology of cancer-related psychiatric disorders is multifactorial and is related to several neuropsychological and neurobiological factors. Specifically, the production of cytokines associated with cancer appears to play a role in the development of depression. Tumours trigger an inflammatory response that leads to the release of pro-inflammatory cytokines. These cytokines influence central nervous system function and disrupt the regulation of the HPA axis, contributing to psychological symptoms such as depression, fatigue, sleep disturbances, and appetite loss.

Moreover, psychiatric symptoms in cancer patients are often accompanied by neuropsychological alterations including deficits in memory, executive function, and attention. Compared to other individuals with psychiatric disorders, cancer patients may experience more severe cognitive impairments which can be exacerbated by cancer treatments, including surgery, chemotherapy, and radiotherapy. These treatments stimulate cytokine production by nearby non-cancerous cells and immune cells activated in response to treatment-induced cell death, thereby driving systemic inflammation.

Cancer profoundly affects not only patients but also their families, who often bear the emotional and caregiving burden. Being close to a loved one with cancer can lead to significant psychological distress, including anxiety and depression, among family members and caregivers. The ripple effects of this burden underscore the need for a holistic approach to mental health in oncology.

Given the background presented so far, identifying and managing psychiatric comorbidities in oncological patients and their families is crucial. This multifaceted interplay between cancer and psychiatric disorders necessitates a comprehensive, interdisciplinary approach to understanding, diagnosing, and treating these conditions effectively.

DETAILED DESCRIPTION:
Cancer is among the leading causes of morbidity and mortality worldwide, profoundly affecting patients' lives at every level. While considerable advances have been made in understanding and treating the biological aspects of cancer, its psychological and psychiatric impacts remain a major concern. Psychiatric disorders, including depression, anxiety, post-traumatic stress disorder (PTSD), and adjustment disorders, are frequently observed in cancer patients. These disorders are not only common but also underdiagnosed, as their symptoms are often misinterpreted as normal emotional reactions to the illness. This misperception undermines the recognition of significant psychiatric conditions that require targeted interventions. Still, psychiatric disorders in cancer patients are not merely secondary complications but may actively contribute to poor oncological outcomes. For instance, stress and depression can directly affect tumour biology through neuroendocrine and immune mechanisms, including increased inflammatory responses and dysregulated cortisol levels, via the chronic activation of the Hypothalamic-Pituitary-Adrenal axis (HPA). Indirectly, psychiatric symptoms can impair treatment adherence and lead to lifestyle choices that increase the risk of recurrence, such as poor nutrition, lack of physical activity, or substance use.

The pathophysiology of cancer-related psychiatric disorders is multifactorial and is related to several neuropsychological and neurobiological factors. Specifically, dysregulation of biology in cancer patients might confer greater vulnerability to psychiatric disorders. The production of cytokines associated with cancer appears to play a role in the development of depression. Tumours trigger an inflammatory response that leads to the release of pro-inflammatory cytokines, including IL-6, TNF-α, CRP, and IL-1ra. These cytokines influence central nervous system function and disrupt the regulation of the HPA axis, contributing to psychological symptoms such as depression, fatigue, sleep disturbances, and appetite loss. Since tumour-related inflammation emerges early in the progression of cancer, depression and other psychological symptoms might manifest as initial indicators of the disease.

Moreover, psychiatric symptoms in cancer patients are often accompanied by neuropsychological alterations including deficits in memory, executive function, and attention. Compared to other individuals with psychiatric disorders, cancer patients may experience more severe cognitive impairments which can be exacerbated by cancer treatments, including surgery, chemotherapy, and radiotherapy. These treatments stimulate cytokine production by nearby non-cancerous cells and immune cells activated in response to treatment-induced cell death, thereby driving systemic inflammation.

Cancer profoundly affects not only patients but also their families, who often bear the emotional and caregiving burden. Being close to a loved one with cancer can lead to significant psychological distress, including anxiety and depression, among family members and caregivers. The ripple effects of this burden underscore the need for a holistic approach to mental health in oncology.

Given the background presented so far, identifying and managing psychiatric comorbidities in oncological patients is crucial. However, there are several difficulties in assessing these patients. First, there is a need to better understand the psychopathology behind cancer. Frequently, symptoms like depression and anxiety are conceived as normal reactions to cancer, whereas cancer can trigger severe syndromes, which are frequently overlooked. Second, studies related to common biological patterns linking cancer and psychiatric disorders are poorly investigated. Furthermore, there is a lack of studies that assess the effectiveness and safety of pharmacological and non-pharmacological treatments in these patients.

Family members of cancer patients experience significant emotional and psychological strain, yet their psychiatric symptoms are often overlooked. The biological underpinnings of these symptoms in caregivers, as well as effective treatments tailored to this population, are under-researched. Addressing the mental health needs of families is essential to improving overall care outcomes in oncology.

This multifaceted interplay between cancer and psychiatric disorders necessitates a comprehensive, interdisciplinary approach to understanding, diagnosing, and treating these conditions effectively.

ELIGIBILITY:
Inclusion Criteria:

* For cases: any subject affected by cancer with a comorbid psychiatric disorder (further defined as "cases") or any first-degree relative of a subject of a "case" (i.e., i.e. a fist-degree relative of a subject affected by cancer and a psychiatric disorder). These first-degree relatives will be defined as "cases-rel".
* For controls: a) Subjects with cancer who will undergo a consultation in the Clinical and Emergency Psychiatry Unit of the Fondazione Policlinico Universitario Agostino Gemelli IRCCS but who do not show any psychiatric symptoms (further defined as "oncology-controls"); b) subjects without cancer who will undergo a psychiatric evaluation in the Clinical and Emergency Psychiatry Unit and present psychiatric symptoms (further defined as "psy-controls"); c) Subjects without cancer and with any suspected psychiatric disorder who will undergo a psychiatric evaluation in the Clinical and Emergency Psychiatry Unit and who are not diagnosed with any relevant psychiatric symptoms after the evaluation (further defined as "healthy controls"); d) First-degree relatives of "oncology-controls", "psy-controls" and "healthy controls" (further defined as "control-rel").
* Age between 18 and 75 years.
* Capability of providing written informed consent.

Exclusion Criteria:

* Severe cognitive impairment or inability to provide written informed consent.
* Severe unstable neurological disorders, such as traumatic brain injury, Alzheimer's Disease or dementia.
* Inability to perform psychiatric or neuropsychological evaluations.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants will be recruited in the Clinical and Emergency Psychiatry Unit of the Fondazione Policlinico Universitario Agostino Gemelli IRCCS. The Clinical and Emergency Psychiatry Unit and provides outpatient psychiatric assessments and consultations in inpatients wards and day hospitals of the aforementioned institution. Subjects will undergo a first psychiatric evaluation by a clinician of the aforementioned unit. Then, the subject will be assigned to one of the study groups (see above).
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2026-01-30 (Estimated); Primary Completion 2036-01-29 (Estimated); Study Completion 2036-01-29 (Estimated)

PRIMARY OUTCOMES:
Psychiatric differences | January 2026 - January 2035
  Evaluate psychiatric differences among cases and controls over the time

SECONDARY OUTCOMES:
Demographic characteristics course over time | January 2026 - January 2035
  Evaluate differences of certain demographical characteristics among cases and controls over time
Medical characteristics course over time | January 2026 - January 2035
  Evaluate presence/absence of certain medical characteristics among cases and controls over time
Biological characteristics course over time | January 2026 - January 2035
  Evaluate presence/absence of certain biological characteristics among cases and controls over time
Neuropsychological characteristics course over time | January 2026 - January 2035
  Evaluate presence/absence of certain neuropsychological characteristics among cases and controls over time
Differences in psychiatric symptoms in subjects under different medications | January 2026 - January 2035
  Evaluate differences in presence/absence of certain psychiatric symptoms among subjects under certain medications and their course over time
Differences in psychiatric rating scales in subjects under different medications | January 2026 - January 2035
  Evaluate differences in scores of psychiatric rating scales among subjects under certain medications and their course over time
Differences in biological characteristics and their course over time | January 2026 - January 2035
  Evaluate differences among cases and controls over time in levels of C-reactive protein, erythrocyte sedimentation rate, interleukines, vitamin D, folate, vitamin B12, iron, ferritin, transferrin, total iron-binding capacity, glucose, insulin, glycated hemoglobin, triglycerides, cholesterol , apolipoproteins, aspartate aminotransferase, alanine aminotransferase, alkaline phosphatase, gamma-glutamyl transferase, bilirubin, glomerular filtration rate, uric acid, sodium, potassium, chloride, calcium, magnesium, phosphorus, cortisol, adrenocorticotropic hormone, prothrombin time, activated partial thromboplastin time, international normalized ratio, fibrinogen, white blood cell count, red blood cell count, hemoglobin, platelet count, mean corpuscular volume, mean corpuscular hemoglobin, mean corpuscular hemoglobin concentration, red cell distribution width, neutrophil-to-lymphocyte ratio, and albumin and prealbumin levels.
Biological differences in subjects under different medications | January 2026 - January 2035
  Evaluate differences and their course over time of the following biological parameters: C-reactive protein, erythrocyte sedimentation rate, interleukines, vitamin D, folate, vitamin B12, iron, ferritin, transferrin, total iron-binding capacity, glucose, insulin, glycated hemoglobin, triglycerides, cholesterol , apolipoproteins, transaminases, alkaline phosphatase, bilirubin, glomerular filtration rate, uric acid, sodium, potassium, chloride, calcium, magnesium, phosphorus, cortisol, adrenocorticotropic hormone, prothrombin time, activated partial thromboplastin time, international normalized ratio, fibrinogen, white blood cell count, red blood cell count, hemoglobin, platelet count, neutrophil-to-lymphocyte ratio, and albumin and prealbumin levels.
  Comparisons will be made in subjects undergoing different medicatiosns such as antidepressants, mood stabilizers, antipsychotics, benzodiazepines, stimulants.
Side effects | January 2026 - January 2035
  Compare rates of side effects related to different classes of pharmacological treatments.
Correlations between biology and neuropsychology and illness burden | January 2026 - January 2035
  Correlate alterations of neuropsychology and biological markers (inflammatory cytokines and blood cells count,) with severity of psychiatric symptoms at T0 and the evolution of these relationships over time.